CLINICAL TRIAL: NCT02390232
Title: Prospective Cohort Assessing the Role of the Genotoxin Colibactin From Escherichia Coli B2 in the Genesis of NASH
Acronym: Coli-NASH
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/14/7319
Record Dates: First submitted 2015-02-25; First posted 2015-03-17 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: gut microbiota; Non Alcoholic Steato Hepatitis; Steatohepatitis; Escherichia coli; colibactin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Escherichia coli Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — feces, liver, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NAFLD with simple steatosis: Patients with NAFLD with simple steatosis: collection of stools, blood sample and liver biopsy
  Interventions: Biological: liver biopsy; Biological: collection of stools; Biological: blood sample
- NAFLD with steatohepatitis: Patients with NAFLD with steatohepatitis: collection of stools, blood and liver biopsy
  Interventions: Biological: liver biopsy; Biological: collection of stools; Biological: blood sample

INTERVENTIONS:
Biological: liver biopsy — A small needle is inserted into the liver to collect a tissue sample
Biological: collection of stools — collection of stools
Biological: blood sample — collection of blood sample

SUMMARY:
In a population of patients with Non Alcoholic Fatty Liver Disease (NAFLD), the investigators will compare the composition of the gut microbiota from patients with simple steatosis with that with steatohepatitis.

The purpose of this study is to determine if the pathogenic Escherichia Coli to the B2 group and producing the genotoxin colibactin is a factor for developing NASH.

DETAILED DESCRIPTION:
Gut microbiota composition is now linked to the onset of obesity, metabolic disorders, and Non Alcoholic Fatty Liver Disease . While simple steatosis has benign prognosis, steatohepatitis (NASH) leads to cirrhosis and hepatocarcinoma and increases cardiovascular and cancer- related mortality. Some Escherichia coli (E. coli) belonging to the B2 phylogenetic group are involved in many diseases. Those producing the genotoxin colibactin are in addition known to induce a chronic alteration of intestinal permeability, one of the major factors leading to NASH.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD
* indication of liver biopsy

Exclusion Criteria:

* presence of any other cause of liver or steatosis
* alcohol consumption exceeding 30 g / day for a men and 20 g / day for a woman
* a history of decompensated cirrhosis
* treatment with prebiotics, probiotics or antibiotics in the month prior to inclusion
* chronic gastrointestinal disease or history of gastrointestinal surgery
* pregnancy or breastfeeding
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non Alcoholic Fatty Liver Disease
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
composition of the gut microbiota between two groups, and prevalence of the Escherichia Coli belonging to the B2 group and producing the genotoxin colibactin. | 1 day
  compare the composition of the gut microbiota between patients with simple steatosis with steatohepatitis, and determinate the prevalence of the Escherichia Coli belonging to the B2 group and producing the genotoxin colibactin.

SECONDARY OUTCOMES:
differences between the two groups | 1 day
  highlight other differences between the two cohort
determine wether bacteria, in particular escherichia Coli can translocate and reach steatohepatitis patients liver | 1 day
  determine if bacteria, in particular escherichia Coli can translocate and reach steatohepatitis patients liver
Exploration of a biomarker of fibrosis from blood microbiota in NAFLD patients | 1 day
  Determination of bacterial translocation assay PCR 16S bacterial gene in blood and sequence and analyse the microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Maeva Guillaume, Doctor, Principal Investigator — CHU de Toulouse, hôpital Purpan
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smati S, Polizzi A, Fougerat A, Ellero-Simatos S, Blum Y, Lippi Y, Regnier M, Laroyenne A, Huillet M, Arif M, Zhang C, Lasserre F, Marrot A, Al Saati T, Wan J, Sommer C, Naylies C, Batut A, Lukowicz C, Fougeray T, Tramunt B, Dubot P, Smith L, Bertrand-Michel J, Hennuyer N, Pradere JP, Staels B, Burcelin R, Lenfant F, Arnal JF, Levade T, Gamet-Payrastre L, Lagarrigue S, Loiseau N, Lotersztajn S, Postic C, Wahli W, Bureau C, Guillaume M, Mardinoglu A, Montagner A, Gourdy P, Guillou H. Integrative study of diet-induced mouse models of NAFLD identifies PPARalpha as a sexually dimorphic drug target. Gut. 2022 Apr;71(4):807-821. doi: 10.1136/gutjnl-2020-323323. Epub 2021 Apr 26. PMID 33903148